CLINICAL TRIAL: NCT05848934
Title: Evaluation and Prognosis of Cerebrovascular and Neurological Health Status in Patients With Coronary Heart Disease After Treatment
Brief Title: Research on the Relationship Between Cognitive Function Changes and Cerebrovascular Health in Patients With Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Collaborators: Xi'an Jiaotong University (Other); Yuncheng First Hospital (Unknown)
Responsible Party: Principal Investigator, Qianyan Liu, Principal Investgator, Nanjing University of Traditional Chinese Medicine
Other Study IDs: 82071993-1
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Coronary Heart Disease; Image
Keywords: Coronary Heart Disease; MRI Imaging; Neuropsychological assessment
MeSH Terms: conditions — Coronary Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CAD（coronary heart disease ）surgical treatment
  Interventions: Device: magnetic resonance image; Diagnostic Test: Neuropsychological scale
- CAD（coronary heart disease ）conservative treatment
  Interventions: Device: magnetic resonance image; Diagnostic Test: Neuropsychological scale
- HC （Healthy controls）
  Interventions: Device: magnetic resonance image; Diagnostic Test: Neuropsychological scale

INTERVENTIONS:
Device: magnetic resonance image — Imaging data were collected in a strong magnetic field
Diagnostic Test: Neuropsychological scale — Multi dimensional neuropsychological test

SUMMARY:
The purpose of this study is to elucidate the imaging mechanisms of cognitive function changes in patients with coronary heart disease before and after surgery or conservative treatment, and to evaluate and predict the postoperative neurological function recovery and cerebrovascular health level of patients by combining serum markers and patient cardiovascular health evaluation indicators.

DETAILED DESCRIPTION:
The focus of this study is to elucidate the impact of coronary heart disease on the morphology and cognitive changes of cerebral blood vessels in patients. Record imaging data, neuropsychological cognitive scales, serum markers, adverse cardiac events, and patient evaluation indicators before and after clinical treatment and follow-up period, and explore relevant factors affecting changes in cerebrovascular morphology and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed coronary heart disease or risk of coronary heart disease through clinical testing
* Conscious and capable of completing neuropsychological scales

Exclusion Criteria:

* Patients with other serious heart diseases (such as aortic aneurysm)
* People with uncontrolled hypertension or diabetes
* There are contraindications to MRI examination (there are metal implants in the body, such as cardiac pacemakers, metal dentures, artificial joints, non paramagnetism stents, etc.; there is claustrophobia)
* Have a history of severe stroke, epilepsy, traumatic brain injury, and transient ischemic events
* Existence of neurological and mental disorders (schizophrenia, depression, etc.), post-traumatic stress disorder, obsessive-compulsive disorder, multiple sclerosis, amyotrophic lateral sclerosis, etc
* Have a history of alcohol or drug abuse
* Those with significant organ dysfunction such as lung, liver, and kidney;
* Patients with tumor, infectious diseases, blood system disease and immune system disease;
* Currently participating in other clinical studies at the same time.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the patients of CAD（coronary heart disease ）surgical treatment group and CAD（coronary heart disease ）conservative treatment group are in-patients and out-patients in the cardiac surgery department from the research center. The subjects of healthy control group are recruited from community.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of brain volume before and after treatment | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of brain volume (mm3) are evaluated by structural 3DT1 weighted MRI. Freesurfer software is used to get the measured value of the volume.
Change of cerebrovascular morphology before and after treatment | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of Cerebral vessel density, caliber and tortuosity, brain white matter hyperintensity lesion count
Change of brain function connectivity before and after operation | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of brain functional connectivity intensity are evaluated by rest stage functional MRI. DPABI software based on MATLAB is used to get the measured the matrix value of functional connectivity.

SECONDARY OUTCOMES:
Change of serum marker concentration before and after operation | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of serum marker concentration is evaluated by inflammatory cytokine.
Change of plasma marker concentration before and after operation | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of plasma marker concentration is evaluated by neurofilament light chain(NFL) protein extracted from plasma.
Change of cardiovascular risk factors before and after operation | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of cardiovascular risk factors is evaluated by blood routine and patients' living habits
Change of executive functions before and after operation evaluated by Trail-Making Test Part A | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of executive functions are first evaluated by Trail-Making Test Part A test. The minimum value is 0 , and the maximum value is 30. This test has no clear maximum and minimum values. If the test completion time exceeds 79 seconds, it means the outcome is abnormal. The higher scores mean a worse outcome.
Change of working memory before and after operation evaluated by Forward Digit Span | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of working memory is first evaluated by Forward Digit Span. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 7.75±1.47. The higher scores mean a better outcome.
Change of working memory before and after operation evaluated by Backward Digit Span | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of working memory is second evaluated by Backward Digit Span. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 5.36±1.91. The higher scores mean a better outcome.
Change of executive functions before and after operation evaluated by Trail-Making Test Part B | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of executive functions are first evaluated by Trail-Making Test Part B test. The minimum value is 0 , and the maximum value is 30. This test has no clear maximum and minimum values. If the test completion time exceeds 79 seconds, it means the outcome is abnormal. The higher scores mean a worse outcome.It is a supplement to Trail-Making Test Part A, which is optional for patients who are not familiar with the English alphabetical order
Change of executive functions before and after operation evaluated by Digit Symbol Coding score | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of executive functions are second evaluated by Digit Symbol Coding score. The minimum value is 0 , and the maximum value is not clear. The normal range of results is 56.53 ± 20.17. The higher scores mean a better outcome.
Change of episodic memory functions before and after operation evaluated by Auditory Verbal Learning test | before operation; 3-10 Days after operation; 1 month; 6-12months
  The change of episodic memory are evaluated by Auditory Verbal Learning test(AVLT-H).

CONTACTS AND LOCATIONS:
Overall Officials: Nengrui Guo, Principal Investigator — Yuncheng First Hospital
Locations (1):
- Yuncheng First Hospital, Yuncheng, Shanxi, China